CLINICAL TRIAL: NCT02525796
Title: Evaluating Alternative Medical Therapies in Primary Hyperparathyroidism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anand Vaidya, Assistant Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 107407
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Eplerenone; Amiloride; Cinacalcet

STUDY DESIGN:
Intervention Model Description: 3-parallel-armed double-blinded randomized controlled trial wherein monotherapy of eplerenone or amiloride or placebo administered for 4 weeks. After weeks, an open-label extension addition of cinacalcet to all 3 arms conducted for 2 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo + Cinacalcet (Placebo Comparator): Patients with primary hyperparathyroidism will receive placebo for 4 weeks followed by the addition of cinacalcet for 2 weeks
  Interventions: Drug: Placebo; Drug: Cinacalcet
- Amiloride + Cinacalcet (Active Comparator): Patients with primary hyperparathyroidism will receive amiloride for 4 weeks followed by the addition of cinacalcet for 2 weeks
  Interventions: Drug: amiloride; Drug: Cinacalcet
- Eplerenone + Cinacalcet (Experimental): Patients with primary hyperparathyroidism will receive eplerenone for 4 weeks followed by the addition of cinacalcet for 2 weeks
  Interventions: Drug: eplerenone; Drug: Cinacalcet

INTERVENTIONS:
Drug: eplerenone — eplerenone, titrated up to a maximum of 50mg BID
  Arms: Eplerenone + Cinacalcet
Drug: amiloride — amiloride, titrated up to a maximum of 10mg BID
  Arms: Amiloride + Cinacalcet
Drug: Placebo
  Arms: Placebo + Cinacalcet
Drug: Cinacalcet — Cinacalcet, as add-on therapy in addition to eplerenone/amiloride/placebo, titrated up to a maximum of 30mg BID

SUMMARY:
This study will evaluate whether blocking the mineralocorticoid receptor, alone, or in combination with the calcimimetic cinacalcet, can lower parathyroid hormone and calcium levels in primary hyperparathyroidism.

DETAILED DESCRIPTION:
To conduct a double-blinded, placebo-controlled, randomized intervention study to investigate whether mineralocorticoid receptor (MR) antagonism, alone or in combination with cinacalcet, is an effective therapy for primary hyperparathyroidism (P-HPTH).

Hypothesis: MR antagonism, as a monotherapy or in combination with a calcimimetic, is a mechanism to lower parathyroid hormone (PTH) in primary hyperparathyroidism (P-HPTH).

Study Design: Sixty subjects with P-HPTH will be enrolled to randomly receive eplerenone (a potassium-sparing diuretic that directly blocks the MR), amiloride (a potassium-sparing diuretic that does not directly block the MR), or placebo for 4 weeks. Thereafter, all subjects will receive cinacalcet therapy (a calcimimetic that lowers PTH) in addition to their randomized intervention for an additional 2 weeks.

Anticipated Results: In this proof-of-concept study, eplerenone therapy will lower PTH, serum calcium, and markers of bone resorption in P-HPTH, when compared to placebo. The PTH response to amiloride will resemble that of placebo, suggesting that the eplerenone mediated reductions in PTH are specific to interactions with the MR. Combination therapy with eplerenone + cinacalcet will result in additive or synergistic reductions in PTH, when compared to placebo + cinacalcet or placebo + amiloride.

Implications: MR antagonism (alone or in combination with cinacalcet) may be a mechanism to lower PTH and calcium in P-HPTH, thereby identifying a new potential option in the limited medical therapies for P-HPTH.

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosis of active P-HPTH (Serum calcium > upper limit of reference range and serum PTH > ULRR; or Serum Calcium > ULRR AND serum PTH > 30 pg/mL; or Serum Calcium within 0.2 mg/dL of the ULRR and PTH>ULRR).
* negative pregnancy test in women aged 18-45

Exclusion Criteria:

* estimated glomerular filtration rate < 60mL/min/1,73m2
* serum potassium > 5.0 mmol/L
* age <18 or >80 years
* diabetes that is not well controlled (HbA1c>8%)\
* liver failure
* heart failure
* history of myocardial infarction or stroke
* active use of lithium
* active chronic inflammatory conditions (such as inflammatory bowel disease, rheumatoid arthritis, sarcoidosis)
* initiation within 3 months of bisphosphonates or cinacalcet
* need for imminent parathyroidectomy (within the next 6-8 weeks) as determined by their endocrinologist or surgeon
* absolute serum calcium >13.0 mg/dL
* positive pregnancy test on any of the study visits for women ages 18-45.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Vaidya, MD MMSc, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with interested investigators upon request 1 year after the study is completed. Investigators may request IPD by contacting the PI and proposing a data analysis plan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment (n=69), participants underwent medication washout to eliminate interference with renin-angiotensin-aldosterone system measurements. ACE inhibitors, ARBs, ENaC inhibitors, and MR antagonists were stopped for 2 weeks and BP controlled with alternative agents, if needed. During washout, 28 participants were withdrawn, thus the number of participants at the time of randomization to monotherapy was 41. 36 of 41 completed 4wks and began the cinacalcet open-label phase.
Groups:
- Eplerenone: Patients with primary hyperparathyroidism will receive maximally-tolerated, double-blinded, eplerenone monotherapy for 4 weeks, followed by an open-label extension wherein maximally-tolerated cinacalcet therapy will be added to eplerenone for 2 weeks.
- Amiloride: Patients with primary hyperparathyroidism will receive maximally-tolerated, double-blinded, amiloride monotherapy for 4 weeks, , followed by an open-label extension wherein maximally-tolerated cinacalcet therapy will be added to amiloride for 2 weeks.
- Placebo: Patients with primary hyperparathyroidism will receive maximally-tolerated, double-blinded, placebo monotherapy for 4 weeks, followed by an open-label extension wherein maximally-tolerated cinacalcet therapy will be added to placebo for 2 weeks.
Period: Randomization to Monotherapy for 4 Weeks
Arm/Group | Eplerenone | Amiloride | Placebo
Started | 14 | 14 | 13
Completed | 12 | 12 | 12
Not Completed | 2 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Open-label Addition of Cinacalcet
Arm/Group | Eplerenone | Amiloride | Placebo
Started | 12 | 12 | 12
Open-label Cinacalcet | 12 (Eplerenone+Cinacalcet) | 12 (Amiloride+Cincalcet) | 12 (Placebo+Cinacalcet)
Completed | 8 | 10 | 9
Not Completed | 4 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Adverse Event | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patient with primary hyperparathyroidism
Groups:
- Eplerenone: Patients with primary hyperparathyroidism will receive maximally-tolerated eplerenone for 4 weeks
- Amiloride: Patients with primary hyperparathyroidism will receive maximally-tolerated amiloride for 4 weeks
- Placebo: Patients with primary hyperparathyroidism will receive placebo for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Eplerenone | Amiloride | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 13 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 3 | 19
  >=65 years | 7 | 5 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 61 (9) | 69 (10) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 11 | 34
  Male | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 1 | 6
  White | 12 | 7 | 12 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 13 | 41
Parathyroid hormone [Mean (Standard Deviation); unit: pg/mL] | 65 (17) | 89 (56) | 66 (26) | 74 (39)
Serum calcium [Mean (Standard Deviation); unit: mg/dL] | 10.4 (0.5) | 10.5 (0.5) | 10.4 (0.6) | 10.5 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Parathyroid Hormone Levels
Description: Change in circulating PTH levels before and after 4 weeks of double-blinded intervention when compared to placebo
Time Frame: Change in circulating PTH levels before and after 4 weeks of double-blinded monotherapy intervention when compared to placebo (PTH at 4 weeks minus PTH at baseline)
Population: Number of participants who completed the 4 week double-blinded monotherapy intervention
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Eplerenone: Patients with primary hyperparathyroidism will receive maximally-tolerated eplerenone monotherapy for 4 weeks
- Amiloride: Patients with primary hyperparathyroidism will receive maximally-tolerated amiloride monotherapy for 4 weeks
- Placebo: Patients with primary hyperparathyroidism will receive placebo monotherapy for 4 weeks
Arm/Group | Eplerenone | Amiloride | Placebo
Number analyzed (Participants) | 12 | 12 | 12
pg/mL | 4.0 [-10.4 to 10.4] | -3.7 [-11.4 to 8.7] | 0.8 [-3.6 to 8.3]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; ANOVA comparing the change in PTH over 4 weeks between eplerenone monotherapy and placebo; Test type: Superiority; p = 0.84, ANOVA; Median Difference (Net) = 3.2
Statistical Analysis 2: Comparison: Amiloride vs Placebo; ANOVA comparing the change in PTH over 4 weeks between amiloride monotherapy and placebo; Test type: Superiority; p = 0.54, ANOVA; Median Difference (Net) = 4.5
Statistical Analysis 3: Comparison: Eplerenone vs Amiloride; ANOVA comparing the change in PTH over 4 weeks between eplerenone monotherapy and amiloride monotherapy; Test type: Superiority; p = 0.58, ANOVA; Median Difference (Net) = 7.6

2. Secondary Outcome: Change in Calcium Levels
Description: Change in serum calcium levels before and after intervention when compared to placebo
Time Frame: Change in serum calcium levels before and after 4 weeks of double-blinded monotherapy intervention when compared to placebo (calcium at 4 weeks minus calcium at baseline)
Population: patients with primary hyperparathyroidism receiving double-blinded monotherapy for 4 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Eplerenone | Amiloride | Placebo
Number analyzed (Participants) | 12 | 12 | 12
mg/dL | 0.1 [-0.1 to 03] | 0.0 [-0.3 to 0.1] | 0.1 [-0.1 to 0.4]
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; ANOVA comparing the change in serum calcium over 4 weeks between eplerenone monotherapy and placebo; Test type: Superiority; p = 0.82, ANOVA; Median Difference (Net) = 0
Statistical Analysis 2: Comparison: Amiloride vs Placebo; ANOVA comparing the change in serum calcium over 4 weeks between amiloride monotherapy and placebo; Test type: Superiority; p = 0.21, ANOVA; Median Difference (Net) = 0.1
Statistical Analysis 3: Comparison: Eplerenone vs Amiloride; ANOVA comparing the change in serum calcium over 4 weeks between eplerenone monotherapy and amiloride monotherapy; Test type: Superiority; p = 0.12, ANOVA; Median Difference (Net) = 0.1

ADVERSE EVENTS:
Time Frame: Over the course of the entire study, including the 4 week randomization to monotherapy (eplerenone vs amiloride vs placebo) and the 2 week open-label addition of cinacalcet (6 weeks in total).
Description: same as clinicaltrials.gov
Groups:
- Eplerenone + Cinacalcet; Amiloride + Cinacalcet; Placebo + Cinacalcet: Open-label cinacalcet added for 2 weeks
Arm/Group | Eplerenone | Amiloride | Placebo | Eplerenone + Cinacalcet | Amiloride + Cinacalcet | Placebo + Cinacalcet
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14 | 1/13 | 2/12 | 2/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone (N=14) | Amiloride (N=14) | Placebo (N=13) | Eplerenone + Cinacalcet (N=12) | Amiloride + Cinacalcet (N=12) | Placebo + Cinacalcet (N=12)
low egfr (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
hyperkalemia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
hypocalcemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — low serum calcium
low blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — blood pressure below target range

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02525796/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT02525796/SAP_001.pdf